CLINICAL TRIAL: NCT04378218
Title: Cardiovascular Effects of High Intensity Interval Training in Individuals With Paraplegia
Acronym: HIIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kristin L. Garlanger, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-004972
Record Dates: First submitted 2019-11-07; First posted 2020-05-07 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Paraplegia, Spinal; Spinal Cord Trauma
Keywords: HIIT
MeSH Terms: conditions — Paraplegia; Spinal Cord Injuries | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Pre-post trial, observational, feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIIT Intervention (Experimental)
  Interventions: Behavioral: High Intensity Interval Training (HIIT)

INTERVENTIONS:
Behavioral: High Intensity Interval Training (HIIT) — A 16 week, 3 sessions per week HIIT program from the subject's personal wheelchair, positioned near an adjustable table with an arm-ergometer affixed.

SUMMARY:
The study seeks to determine whether high intensity interval training has an effect on cardiovascular parameters in wheelchair users with paraplegia.

DETAILED DESCRIPTION:
The objective of this pilot study is to produce preliminary data testing the feasibility and effectiveness of high intensity interval training (HIIT) on cardiovascular health parameters in individuals with paraplegia. The long term research goal is to determine whether these short term physiologic effects translate to long term reduction in cardiovascular disease and mortality in this high risk population. The rationale for this study is that identifying a well-accepted form of exercise in individuals with paraplegia, which is safe and effective in improving cardiovascular health parameters, would provide an efficient and sustainable evidence-based approach to lowering cardiovascular disease risk. We propose the following two Specific Aims:

Specific Aim #1: Measure cardiovascular changes after a 16-week HIIT program in individuals with paraplegia. Measurements will include oxygen utilization during maximal exercise via VO2max testing (primary outcome measure), body composition via dual energy X-ray absorptiometry, blood lipid panel, C-reactive protein blood test, and glucose utilization via oral glucose tolerance blood test.

Specific Aim #2: Investigate the feasibility, sustainability and acceptance of implementing high-intensity interval training (HIIT) via arm-ergometer as a form of home exercise in individuals with paraplegia. After the personalized training session with the arm-ergometer and the HIIT protocol, each participant will be given an arm-ergometer (also known as arm-cycle) to use within their home to complete three sessions weekly for the entire16 week program. An adjustable table will be provided to allow for height customization of each arm-ergometer, and provide a method for securing the device during exercise. The arm-ergometers allow the subject to complete the exercise intervention from their own wheelchair. Compliance will be monitored via chest strap heart rate monitors. Acceptance of the program will be determined through a pre- and post- training survey Spinal Cord Injury Exercise Self-Efficacy Scale (SCI ESES) and interview with participants.

At the completion of this project, we expect to have determined whether HIIT is an appropriate form of exercise intervention for individuals with paraplegia, effective in improving short-term cardiovascular health parameters within a 16 week home program. We anticipate participants will find HIIT acceptable given the time-efficiency of the protocol, the convenience of using their own wheelchair and the elimination of environmental barriers by performing the program within their home. This study is expected to have a positive impact on cardiovascular health in individuals with paraplegia and foresee this form of exercise being implemented as a standard of care recommendation in the physical activity guidelines for individuals with paraplegia.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury located at or below the seventh thoracic vertebrae
* Manual wheelchair user (primary means of mobility)At least 6 months post-SCI
* At least 18 years of age
* Able to perform a high-intensity exercise program
* Willingness to participate in 16 weeks of an exercise program
* Personal cell phone with the ability to run the Polar Beat application and BlueTooth capabilities

Exclusion Criteria:

* Spinal cord injury at or above the sixth thoracic vertebrae
* Manual wheelchair is not the primary means of mobility (ex. community ambulators, power wheelchair users)
* Any documented or reported health condition that would be contraindicated to a progressive exercise program (active upper limb musculoskeletal injuries, autonomic instability, unstable cardiopulmonary disease such as unstable angina, COPD, etc., or pregnancy).
* Any illness or condition which, based on the research team's assessment, will compromise with the patient's ability to comply with the protocol, patient safety, or the validity of the data collected during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Physical activity | Baseline, Week 8, Week 16
  Change in physical activity, as measured by the Physical Activity Scale for Individuals with Physical Disabilities (PASIPD) survey
Exercise self-efficacy | Baseline, Week 8, Week 16
  Change in exercise self-efficacy, as measured by the SCI Exercise Self-Efficacy Scale (SCI ESES), with changes in individual responses rated as more true indicating more efficacy.
Glucose metabolism | Baseline, Week 8, Week 16
  Changes in metabolism of glucose, as measured by a 120 minute oral glucose tolerance test (OGTT), with lower glucose values indicating more efficient metabolism.
Inflammatory marker | Baseline, Week 8, Week 16
  Changes in measurements of proteins representing inflammatory processes via the C-Reactive Protein blood test, with lower values indicating a state of less cardiovascular risk.
Lipid profile | Baseline, Week 8, Week 16
  Changes in measurements of total cholesterol, triglycerides, HDL, calculated LDL, and non-HDL cholesterol, with lower values (excepting HDL) indicating lower cardiovascular risk.
Oxygen metabolism | Baseline, Week 8, Week 16
  Changes in metabolism of oxygen, as measured by the Graded Exercise Test (GXT), also known as the VO2 Maximum Test, with higher O2 intake values indicating higher aerobic capacity.
Bone mineral density | Baseline, Week 8, Week 16
  Measurement by dual-energy x-ray absorptiometry (DXA) of change in bone mineral content and bone density.
Body composition - body fat mass | Baseline, Week 8, Week 16
  Measurement by dual-energy x-ray absorptiometry (DXA) of change in regional and total body fat mass.
Body composition - lean mass | Baseline, Week 8, Week 16
  Measurement by dual-energy x-ray absorptiometry (DXA) of change in regional and total lean mass.
Body composition - android and gynoid fat percentage | Baseline, Week 8, Week 16
  Measurement by dual-energy x-ray absorptiometry (DXA) of change in regional and total android and gynoid fat percentage.
Body composition - android and gynoid fat ratio | Baseline, Week 8, Week 16
  Measurement by dual-energy x-ray absorptiometry (DXA) of change in regional and total android to gynoid fat ratio.
Body composition - bone mass | Baseline, Week 8, Week 16
  Measurement by dual-energy x-ray absorptiometry (DXA) of change in regional and total bone mass.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin L. Garlanger, D.O., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials